CLINICAL TRIAL: NCT04884490
Title: The Role of High Dose Co-trimoxazole in Severe Covid-19 Patients- a Double Blind Placebo Controlled Randomized Trial
Brief Title: The Role of High Dose Co-trimoxazole in Severe Covid-19 Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Prof. Dr. Shohael Mahmud Arafat, Clinical Professor of Internal Medicine, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BSMMU/2021/4098(A)
Record Dates: First submitted 2021-05-05; First posted 2021-05-13 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: COVID-19 Pneumonia
Keywords: COVID-19, Co-trimoxazole, RCT
MeSH Terms: conditions — COVID-19 | interventions — Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Intervention Model Description: Study design:Single-centre interventional Prospective double-blind placebo controlled randomized trial.
  Study duration: Six months. Place of study: Medicine department (Covid Unit) of Bangabandhu Sheikh Mujib Medical University (BSMMU) Period of Study: Six months following approval of the protocol Sampling technique: Random sampling followed by patients will be assigned in a 1:1 ratio to either oral high dose co-trimoxazole in addition to standard therapy or standard therapy along with placebo
  Sample Size:
  47 in each group
Who Masked: Participant, Care Provider, Investigator
Masking Description: A data sheet (enclosed) will be prepared, for which a short interview of less than 30 minutes will be required. Ethical risks are deemed minimal as standard therapy as well as co-trimoxazole are extensively used treatments and have well-documented efficacy& safety. Placebo will be used here along with standard therapy in the control group. Informed oral and written consent will be taken from the study subjects. Patient will be given packs containing total number of 27 tablets of Co-trimoxazoles or placebo which will be coded by a personnel not involved in the study. Research assistant and investigators will not be aware of the drug. After data collection and entry during analysis decoding will be done.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Eligible patients will be receiving either to oral co-trimoxazole + standard therapy.
  Tab. Co-trimoxazole 960 mg (trimethoprim 160mg + sulphamethoxazole 800mg) thrice (8 hourly) daily for 7 days orally.
  The following treatments are recommended as standard therapy:
  1. Antibiotics for secondary bacterial infection as per institutional guidelines
  2. Supplemental oxygen (to keep saturations between 92% to 96%)
  3. Intravenous hydration (to maintain euvolumia)
  4. Thrombo-prophylaxis as per local guidelines
  5. Paracetamol (oral or I/V 1gram QDS as required or regular)
  6. To consider steroids in appropriate cases.
  7. Nasopharyngeal and throat swab to be sent for RT PCR to detect SARS-CoV-2 (if not already done) and blood culture Tab. Co-trimoxazole 960 mg (trimethoprim 160mg + sulphamethoxazole 800mg) thrice (8 hourly) daily for 7 days orally.
  Interventions: Drug: Co-trimoxazole
- Standard (Placebo Comparator): Standard therapy along with placebo.
  Placebo thrice (8 hourly) for 7 days.
  The following treatments are recommended as standard therapy:
  1. Antibiotics for secondary bacterial infection as per institutional guidelines
  2. Supplemental oxygen (to keep saturations between 92% to 96%)
  3. Intravenous hydration (to maintain euvolumia)
  4. Thrombo-prophylaxis as per local guidelines
  5. Paracetamol (oral or I/V 1gram QDS as required or regular)
  6. To consider steroids in appropriate cases.
  7. Nasopharyngeal and throat swab to be sent for RT PCR to detect SARS-CoV-2 (if not already done) and blood culture
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Co-trimoxazole — Tab. Co-trimoxazole 960 mg (trimethoprim 160mg + sulphamethoxazole 800mg) thrice (8 hourly) daily for 7 days orally.
  Arms: Intervention
Drug: Placebo — Placebo thrice (8 hourly) daily for 7 days orally.
  Arms: Standard

SUMMARY:
Coronavirus Disease 19 (COVID-19) is a worldwide pandemic and a major global health concern which is caused by Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2). The newly emerged Coronavirus disease 2019 (COVID-19), which was first identified in Wuhan, China, has swept through 219 countries, killing a staggering number of people. According to WHO reports, the number of deaths had risen to 3,155,168by March 30, 2021, out of 149,910,744 confirmed cases. In Bangladesh, the outbreak has infected over 745,322confirmed cases, with over 11,053 deaths reported. Though the patient may be asymptomatic or present with mild symptoms, mortality is quite high in the severe form of the disease which often progresses to critical phase presented as Acute Respiratory Distress Syndrome (ARDS). This is due to exaggerated response of immune system to the virus termed as cytokine storm syndrome (CSS). There is currently no effective antiviral therapy for SARS-CoV-2 and supportive care is the mainstay of therapy. As a result we are still searching for a better therapeutic agent which will help in treating Covid-19 cases in terms of mortality, morbidity, oxygen requirement, length of stay in hospital. Co-trimoxazole (composed of one-part Trimethoprim and five parts Sulfamethoxazole)is a sulphur containing anti-folate bactericidal drug which is being used for over 60 years for various indications esp. respiratory tract infections. It is known to have immunomodulatory and anti-inflammatory properties that may help to prevent progression to critical phase and cytokine storm syndrome in severe COVID-19 patients. It acts rapidly when given in high dose due to its better bioavailability and lung penetration. Low cost and a good safety profile can make it an ideal candidate for treatment of COVID -19 in a low resource country like Bangladesh.

Methods and materials:

This interventional double-blind place controlled randomized trial will be conducted in the department of medicine at Bangabandhu Sheikh Mujib Medical University (BSMMU) for a duration of 6 months following approval of this protocol. It will recruit at least 94 consecutive adults (18 years or older) patients with clinically suspected COVID-19 and severe illness as per WHO criteria. After taking informed written consent patients will be randomly assigned in a 1:1 ratio to either oral high dose co-trimoxazole in addition to standard therapy or placebo along with standard therapy. Baseline characteristics, changes in the physiological and biochemical parameters like (SpO2/FiO2 ratio, respiratory rate, body temperature and C - reactive protein), length of hospital stay, side effects of drugs, requirement for ventilatory support (non-invasive and invasive ventilation) and 28- day mortality between the two groups will be compared. Data will be collected from case record forms, anonymised and stored securely in a secure online web based portal. Statistical analysis will be performed using t-test or Mann -Whitney U test or Wilcoxon signed rank test for continuous variables and Chi- square test or Fisher's exact test for categorical variables. Survival will be assessed by the Kaplan-Meier method. Comparisons between two groups will be performed using the log-rank test. A p-value of < 0.05 will be considered to be significant. The statistical software SPSS version 25 will be used for the analysis.

Conclusion If the results from this clinical trial demonstrate the beneficial effects of high co-trimoxazole in patients with severe COVID-19 it could help to reduce the need for respiratory support for thousands of patients, saving valuable lives and decrease the burden of healthcare system in countries with limited resources.

DETAILED DESCRIPTION:
The newly emerged Coronavirus disease 2019 (COVID-19), which was first identified in Wuhan, China, has swept through 219 countries, killing a staggering number of people. The World Health Organization (WHO) has declared the deadly outbreak a pandemic, with far-reaching consequences for all people. According to WHO reports, the number of deaths had risen to 3,155,168by March 30, 2021, out of 149,910,744 confirmed cases.

The pathogen for COVID-19 has been described as the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), a new beta-coronavirus. Following the outbreaks of the severe acute respiratory syndrome (SARS) and Middle East respiratory syndrome (MERS) coronaviruses in 2003 and 2012, respectively, this strain has been the third most deadly pathogenic human coronavirus. In Bangladesh, the outbreak has infected over 745,322confirmed cases, with over 11,053 deaths reported.

COVID-19 is spread from person to person through respiratory droplets. The disease is characterized by respiratory symptoms, the most common of which are fever, fatigue, myalgia, dry cough, and dyspnea.

People with co-morbidities such as diabetes, cardiovascular and cerebrovascular disorders, cancers, and pre-existing lung diseases such as Chronic Obstructive Pulmonary Disease (COPD) have been shown to have a greater risk of developing serious forms of the disease.

Septic shock, coagulation disorders, Acute Respiratory Distress Syndrome (ARDS), multi-organ failure, and even death may occur in people with serious illness.

According to recent research, the SARSCoV-2 envelope spike protein receptor binding domain binds to the angiotensin converting enzyme 2 (ACE2) receptors of the host cells, which are mainly respiratory epithelial cells and alveolar pneumocytes type 2 (AT2).

The virus then induces lysis of the infected cells, causing the release of proinflammatory cytokines such as interleukin (IL) IL1, IL2, IL6, IL 7, interferon gamma, macrophage inflammatory proteins, tumor necrosis factor alpha, and others, initiating the host's inflammatory immune response.

A cytokine storm syndrome (CSS) develops in patients with severe forms of the disease as a result of the host's excessive immune response combined with continued lysis of the infected cells. Damage Associated Molecular Patterns (DAMPs) released after mitochondrial injury in host cells stimulate Formyl Peptide Receptors (FPRs) on the outer surface of neutrophils and monocytes' cell membranes, causing their recruitment to the lungs. FPRs cause the release of Reactive Oxygen Species (ROS) in the tissue when stimulated, which leads to the release of even more cytokines.

This causes extensive tissue damage, causing mild respiratory symptoms like dry cough and fever to quickly progress into Acute Respiratory Distress Syndrome, followed by multiple organ failure in susceptible patients.

A large, randomized clinical trial involving more than 6400 hospitalized patients with Covid-19 showed that dexamethasone significantly reduced 30-day mortality (17% reduction); benefit was limited to patients who required oxygen supplementation and appeared greater in patients receiving mechanical ventilation.10 Consequently, dexamethasone (or potentially other glucocorticoids) is now considered the standard of care for patients with severe Covid-19. Data from a randomized, placebo-controlled trial involving more than 1000 patients with severe Covid-19 showed that the antiviral agent remdesivir reduced time to clinical recovery; the benefit appeared greatest in patients who were receiving supplemental oxygen but were not intubated.11The combination of dexamethasone and remdesivir is increasingly used clinically, but its benefit has not been shown in randomized clinical trials. Tocilizumab, an interleukin-6 inhibitor, did not significantly reduce disease progression.

Therefore in managing severe Covid-19 patients physicians are still searching for better options. The key to managing severe COVID-19 is to prevent this cytokine storm from occurring, as well as to ensure that there are no secondary bacterial infections in the patient's already compromised lungs.

Cotrimoxazole is a common antibiotic used to treat a variety of illnesses, including urinary and respiratory tract infections and opportunistic pneumocystis pneumonia, and toxoplasmosis in HIV/AIDS patients. Being composed of one-part Trimethoprim and five parts Sulfamethoxazole, Cotrimoxazole is a low-cost drug with good effectiveness and a low risk of side effects.

Many studies have shown that Cotrimoxazole has immunomodulatory and anti-inflammatory properties. In the ARROW trial, plasma pro-inflammatory markers like C reactive protein (CRP) and Interleukin 6 were found to be lower in continuous Cotrimoxazole prophylaxis, implying that it has anti-inflammatory and immunomodulatory properties.

Cotrimoxazole has been shown to block FPRs, preventing the recruitment of inflammatory cells, the release of cytokines, and the production of reactive oxygen species (ROS) in damaged tissue.

Cotrimoxazole has also been shown to be effective in lowering pro-inflammatory cytokines such as IL-1, 2, 6, 8, and Tumor Necrosis Factor - α.

This could prevent the clinically serious COVID-19 from progressing to ARDS by preventing the imminent CSS. In addition, the drug is very effective in treating nosocomial and opportunistic infections. This could also help to prevent COVID from progressing to ARDS by avoiding secondary bacterial infection.

A comparative study involving 44 cases, suggested that adding oral Trimethoprim or Cotrimoxazole reduces acute lung injury in patients with severe COVID-19, resulting in decreased need for ventilatory support and improved outcomes. These drugs have no direct antiviral properties, but they may help to prevent ARDS. The positive effects were noticeable within hours of the first dose, owing to their high absorption and lung penetration.

Another study involving 201 patients shown a significant reduction in mortality, intubation rate, length of hospital and critical care stay and inflammatory markers in the patients treated with Cotrimoxazole along with standard treatment compared to the patients treated with standard treatment alone. A higher dose of Cotrimoxazole was used in this study with excellent safety profile.

A randomized control trial with Cotrimoxazole in patients with severe COVID-19 is underway in India and results are awaited (Clinical Trials Registration-India ID CTRI/2020/10/028297).

Another randomized control trial is currently underway led by the author and team where a lower dose of Cotrimoxazole is being used (ClinicalTrials.gov Identifier NCT04470531).20 High dose Co-trimoxazole may have a potential role to play in preventing the exaggerated immune response in the form of cytokine storm syndrome in patients with severe COVID-19 by its anti-inflammatory and immunomodulatory effect.

RATIONALE:

Corona virus disease (COVID-19), caused by SARS-COV2, is a highly transmissible and potentially deadly disease that is currently causing widespread concern in the global public health community. Bangladesh's pandemic situation is also rapidly changing, with positive cases and deaths rising by the day. There is no specific management for this highly lethal viral infection as of yet. However, there are a few medications that may have a positive impact on the patient's recovery. But large randomized controlled trials investigating the efficacy of those agents have not found much promising result specially when it comes to mortality benefit and cost effectiveness. We are still in need of better therapeutics to combat this pandemic situation. Co-trimoxazole is a tried-and-true antibiotic that has been used in clinical practice for over 60 years and is effective against a wide range of bacteria. Co-trimoxazole also has anti-inflammatory, and immunomodulatory properties in addition to its antimicrobial properties. In previous studies Co-trimoxazole has shown to exert anti-cytokine effect by inhibiting interleukin 1, 6 (IL-1, IL-6) and Tumour Necrosis Factor α (TNF α). These are the major cytokines identified in patients with severe COVID-19. Because Cotrimoxazole has been shown to improve clinical outcomes in ARDS patients in some case reports, there is a chance that it may help improve clinical outcomes in COVID-19 patients. The efficacy of a variety of old and new therapeutic agents is being studied all over the world in order to effectively prevent the life-threatening conditions linked to COVID-19. Because of its immunomodulatory effect, low cost, and good safety profile, co-trimoxazole may be an ideal candidate to investigate. If this agent can be found to reduce the oxygen demand or shorten the length of stay in hospital of severe Covid-19 patients it will definitely have a positive impact in the era of pandemic in resource constraint setting like Bangladesh. This research will provide new data on the safety and effectiveness of high-dose Co-trimoxazole, which will hopefully aid in developing an effective treatment protocol for COVID-19 infection.

Research Question:

Is there any beneficial role of high dose co-trimoxazole in patients with severe COVID-19?

Objectives:

General Objectives To compare the role of high dose co-trimoxazole in severeCOVID-19 patients in addition to standard treatment versus standard treatment along with placebo.

Specific Objectives:

To compare the baseline characteristics in severe covid 19 patients.

To compare the length of stay who are treated with high dose co-trimoxazole in addition to standard treatment versus standard treatment along with placebo.

To compare the requirement for oxygen support through high flow nasal cannula who are treated with high dose co-trimoxazole in addition to standard treatment versus standard treatment along with placebo.

To compare the requirement for ventilatory support (non-invasive and invasive ventilation) who are treated with high dose co-trimoxazole in addition to standard treatment versus standard treatment along with placebo.

To assess the mortality in patients with severe COVID-19 who are treated with high dose co-trimoxazole in addition to standard treatment versus standard treatment along with placebo.

To assess the changes in the physiological and biochemical parameters who are treated with co-trimoxazole in addition to standard treatment versus standard treatment along with placebo.

To find out side effects of drugs who are treated with high dose co-trimoxazole in addition to standard treatment versus standard treatment along with placebo.

Methods and procedure:

Study design: Single-centre interventional double-blind placebo controlled randomized trial.

Study duration: Six months. Place of study: Medicine department (Covid Unit) of Bangabandhu Sheikh Mujib Medical University (BSMMU) Period of Study: Six months following approval of the protocol Sampling technique: Random sampling followed by patients will be assigned in a 1:1 ratio to either oral high dose co-trimoxazole in addition to standard therapy or standard therapy along with placebo

Sample Size:

In order to provide reasonable estimates for the power calculation in the current trial, we used data from a recent COVID-19 study that showed decrease in length of stay by about 25%.Based on similar change with the current intervention we estimated that a total of 94 participants would be needed to detect a significant difference with over 90% power. We will conduct an interim power analysis to test these assumptions, using data from 50 individuals, and adjust sample size if power is lower than anticipated.

At least total 94 study population will be included for the study.

ELIGIBILITY:
Inclusion criteria

* Confirmed COVID-19 patients by RT-PCR
* Clinically suspected COVID-19 patients
* Age > 18 years
* Patients requiring oxygen at least> 5L/min up to 15 L/min (by FM/ NRM)to maintain saturation >92% to 96%

NOTE: Clinically suspected COVID-19 = fever (Temperature >37.8 Degree Celsius) + respiratory symptoms + Radiological evidences Exclusion criteria

* Multi-organ failure
* Severe ARDS (requiring HFNC orventilatory support on presentation in the form ofinvasive or non-invasive ventilation)
* Septic Shock
* Severe liver disease
* Acute Heart Failure
* Acute Kidney Injury (where GFR< 15 and plasma-sulfamethoxazoleconcentration cannot be monitored)
* Drug allergy/intolerance to co-trimoxazole / Sulphar sensitivity
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2021-10-14 (Actual); Study Completion 2021-11-14 (Actual)

PRIMARY OUTCOMES:
Length of stay in hospital (in days) | Upto 28 days
  How long the patient needs hospital care

SECONDARY OUTCOMES:
Change in observations after randomization on Day 3 and 7 | Day 3, Day 7
  SpO2/FiO2 ratio
Change in observations after randomization on Day 3 and 7 | Day 3, Day 7
  respiratory rate
Change in observations after randomization on Day 3 and 7 | Day 3, Day 7
  body temperature
Use of High Flow | Day 28
  Requirement of HFNC
ITU requirement | Day 28
  Requirement of NIV ( CPAP/BiPAP)/ Inotrope support/ Dialysis
Use of ventilatory support (invasive or non-invasive ventilation) | Day 28
In-patient mortality | 28 days
  Death in hospital
Side effects of drugs | Day 7
  Rash, Steven- Johnson Syndrome

CONTACTS AND LOCATIONS:
Locations (1):
- Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No